CLINICAL TRIAL: NCT06165029
Title: Intestinal Ultrasound Combined With Visceral Adipose Tissue Predicts Anti-TNF-α Efficacy in Patients With Inflammatory Bowel Disease: a Prospective Study
Brief Title: IUS Combined With VAT Predicts Anti-TNF-α Efficacy in Patients With IBD: a Prospective Study
Status: Recruiting | Type: Observational
Sponsor: The Third Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Li Tian, MD, Li Tian,MD[fu3tianli], The Third Xiangya Hospital of Central South University
Other Study IDs: fu3tianli2
Record Dates: First submitted 2023-11-20; First posted 2023-12-11 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Inflammatory Bowel Diseases; Intestinal Ultrasound; Visceral Adipose Tissue; TNF-α; Predictors
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Inflammatory Bowel Disease (IBD) is a chronic recurrent nonspecific inflammatory disease of the intestinal tract that can involve multiple organs and systems, mainly including Crohn's disease (CD) and ulcerative colitis (UC). Recurrent disease episodes lead to high rates of disability and unemployment, resulting in a heavy social and economic burden. Currently, the main therapeutic agents for IBD include aminosalicylic acid preparations, glucocorticoids, immunosuppressive agents, and biologic agents, e.g. tumor necrosis factor-a (TNF-a) inhibitors, ustekinumab, etc., with TNF-a inhibitors being the most commonly used in IBD.

The latest guidelines and expert consensus on the diagnosis and management of IBD clearly recommend the use of anti-TNF-a agents. However, not all patients are satisfied with the efficacy of anti-TNF-a agents, and studies have shown that up to 33.7% of responders to induction therapy experience secondary loss of response within a year of starting treatment. Patients remain at risk of poor efficacy or treatment failure with these drugs. Therefore, effective prediction of drug efficacy in patients with IBD is an urgent clinical problem, and the discovery of highly sensitive and specific assays that can identify patients most likely to benefit from treatment as well as those most likely to experience a loss of response is important for guiding clinical therapeutic strategies.

Currently, there are no relevant studies at home or abroad on the combination of intestinal ultrasound (IUS) with visceral adipose tissue (VAT) to predict the response to anti-TNF-a therapy in IBD patients. Therefore, the investigators propose for the first time that IUS combined with VAT is used as a method to predict the efficacy of anti-TNF-a therapy in IBD patients and to further guide the development of individualized treatment plans.

DETAILED DESCRIPTION:
Inflammatory Bowel Disease (IBD) is a chronic recurrent nonspecific inflammatory disease of the intestinal tract that can involve multiple organs and systems, mainly including Crohn's disease (CD) and ulcerative colitis (UC). In recent years, the incidence of IBD in newly industrialized countries is rapidly increasing and is becoming younger. Recurrent disease episodes lead to high rates of disability and unemployment, resulting in a heavy social and economic burden. Currently, the main therapeutic agents for IBD include aminosalicylic acid preparations, glucocorticoids, immunosuppressive agents, and biologic agents, e.g. tumor necrosis factor-a (TNF-a) inhibitors, ustekinumab, etc., with TNF-a inhibitors being the most commonly used in IBD.

The latest guidelines and expert consensus on the diagnosis and management of IBD clearly recommend the use of anti-TNF-a agents. However, not all patients are satisfied with the efficacy of anti-TNF-a agents, and studies have shown that up to 33.7% of responders to induction therapy experience secondary loss of response within a year of starting treatment. Patients remain at risk of poor efficacy or treatment failure with these drugs. Therefore, effective prediction of drug efficacy in patients with IBD is an urgent clinical problem, and the discovery of highly sensitive and specific assays that can identify patients most likely to benefit from treatment as well as those most likely to experience a loss of response is important for guiding clinical therapeutic strategies.

In recent years, many studies have begun to focus on the role of intestinal ultrasound (IUS) in the diagnosis of disease, activity, outcome monitoring, and prediction in patients with IBD. As a noninvasive, reproducible, convenient, and inexpensive test, the ability of intestinal ultrasound to be used as a point-of-care ultrasound may dramatically change the frequency of assessing response to therapy and speed up the clinical decision-making process, and guidelines recommend it as a routine test in patients with IBD. Large multicenter studies have shown that most ultrasound markers return to normal within 12 weeks of treatment initiation, and in particular, normalization of bowel thickness (BWT) is highly correlated with clinical response at 12 weeks. Other subsequent studies have also shown that IUS predicts clinical and endoscopic outcomes in patients with IBD, both in UC and CD, but with limitations, and the predictive efficacy of the further-developed bowel ultrasound score is not sufficient for the clinical need.

Visceral adipose tissue (VAT) refers to the white adipose tissue surrounding the viscera, which is mainly divided into omental adipose tissue, mesenteric adipose tissue (MAT), retroperitoneal fat, perigonadal fat, and peripicardial fat. The role of visceral fat in inflammatory diseases has been gradually emphasized, and it has been found that visceral fat has a special secretion function of inflammatory mediators, which can produce a variety of inflammatory factors, such as TNF-α, interleukin- 6 (IL-6), etc., and these factors play an important role in the inflammatory process. A retrospective study analyzed the relationship between VAT levels and infliximab-induced mucosal healing in 97 CD patients, and found that increased VAT levels were independently associated with attenuated mucosal healing. Gu et al. investigated the effect of visceral fat on the response to treatment and the risk of subsequent surgery in patients with IBD who were treated with anti-TNF-α therapy, and found that visceral fat could also serve as a potential predictor of the efficacy of anti-TNF-α therapy.

Currently, there are no relevant studies at home or abroad on the combination of IUS with VAT to predict the response to anti-TNF-a therapy in IBD patients. Therefore, the investigators propose for the first time that IUS combined with VAT is used as a method to predict the efficacy of anti-TNF-a therapy in IBD patients and to further guide the development of individualized treatment plans.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and ≤ 80 years;
* Patients with newly diagnosed or relapsed active IBD;
* Anti-TNF-α monotherapy is proposed to be applied within 1 month after baseline endoscopy;
* No history of abdominal surgery;
* Clearly understand, voluntarily participate in the study, and sign an informed consent form.

Exclusion Criteria:

* Contraindications to anti-TNF-α therapy: allergy, active tuberculosis or other active infections, moderate-to-severe heart failure (NYHA grade III/IV), demyelinating lesions of the nervous system, live vaccination within the last 3 months, pregnancy and lactation;
* Patients with a history of extensive colectomy or recent proposed colectomy, history of colonic mucosal dysplasia;
* Hypersensitivity to the components of SonoVue contrast media.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In the Third Xiangya Hospital of Central South University, patients with newly diagnosed or relapsed IBD treated with anti-TNF-α will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-11-22 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Bowel wall thickness (BWT) | follow-up time of about 54 weeks
  BWT is measured by intestinal ultrasound. BWT≤3mm means that CD is in quiescent, >3mm means CD is active
visceral adipose tissue (VAT) | follow-up time of about 54 weeks
  VAT was obtained from a computed tomography (CT) or magnetic resonance imaging (MRI) scan and measured at the level of the third lumbar vertebra. APP:NIH ImageJ 1.47 (Bathesda, Maryland, America)

CONTACTS AND LOCATIONS:
Overall Officials: Li Tian, Study Chair — The Third Xiangya Hospital of Central South University
Locations (1):
- the Third Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.